CLINICAL TRIAL: NCT02689089
Title: Acceptability and Completion Rates of a New 12 Dose Treatment (3 Month) Compared to the Standard Treatment for Latent TB Infection Treatment
Brief Title: Taima TB: 3HP Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Government of Nunavut (Unknown); Government of Canada (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20160044-01H
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3HP (Other): The interrupted time series design aims to collect data at multiple time points before (standard regimen) and after the introduction of the new 3HP regimen (interruption) to detect if a significant increase in the number of completions has occurred with the new regimen
  Interventions: Drug: 3HP

INTERVENTIONS:
Drug: 3HP — An interrupted time series study design will be used to determine if the introduction of the 3HP regimen will result in more people completing LTBI treatment compared to the standard of 9 months INH twice weekly.
  Other Names: rifapentine, Priftin

SUMMARY:
This phase IV clinical study trial will be conducted among persons who require treatment for LTBI treatment in Iqaluit, Nunavut and Ottawa, Ontario. The primary objective of this study is to compare the proportion of people who complete directly observed prophylactic treatment (DOPT) using the new 3HP regimen to the current standard of 9 months INH.

DETAILED DESCRIPTION:
The treatment of latent tuberculosis infection (LTBI) is a vital component of the overall strategy to reduce TB in a population. Treatment prevents ongoing transmission in communities by preventing the development of active TB disease. The current international standard for the treatment of LTBI is 9 months of Isoniazid (INH). Adherence to this lengthy regimen is one of the greatest impediments to treatment. A recent multi-centered, multi-national randomized control non inferiority trial with approximately 4,000 patients per arm demonstrated that Rifapentine and INH (3HP) given once weekly for a total of 12 doses was as effective as 9 months (252 doses) of daily INH treatment for LTBI.(1) These findings were also replicated in the pediatric population through a pediatric cohort (n=905 eligible participants) nested within the multi-centered international randomized controlled trial with children between ages 2-17 treated with 3HP compared to the INH standard for LTBI.(2) The efficacy and safety of this new regimen have been established. Rifapentine was approved by the United States Food and Drug Administration (FDA) in December of 2014 for the treatment of LTBI but is not yet approved in Canada. The shortened treatment course could increase the number of people who complete LTBI treatment which could lead to a decrease in active TB cases.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-nursing females between the ages of 2-65 years
2. LTBI diagnosis as per Canadian TB Standards using either the Tuberculin Skin Test (TST) or the Interferon Gamma Release Assay (IGRA)
3. Children 2-5 years with negative TSTs who have been in close contact with a case of active TB disease recently
4. Able and willing to provide fully informed consent or parent/guardian able to provide consent

Exclusion Criteria:

1. Suspected or confirmed active TB disease
2. Known allergies to any of the study medications by participant self-report
3. Female participants of childbearing potential who:

   1. have a positive pregnancy test at screening, or
   2. are not willing to use a reliable method of barrier contraception during the study, or
   3. are breastfeeding
4. Unable/unwilling to substitute medications with drug interactions with 3HP, including :

   1. hormonal contraception
   2. HIV infected participants who are on anti-retroviral drugs
   3. other drugs that interact with 3HP (see Table 1)
5. Known contact with an INH or rifampin resistant case
6. Weight < 10 kg
7. Evidence of possible liver damage defined by an aspartate transaminase (AST) level that is more than 3x the upper limit of normal in an asymptomatic patient
8. Porphyria reported by patient
9. Inability to adhere to protocol.
10. Patients may be excluded from the study for other reasons, at the investigator's discretion with detailed documentation.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Completion of treatment | 3 months
  Participants who start and complete treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo G Alvarez, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Institutional approval would be required from research collaborators for the release of this data.

REFERENCES:
- [Background] Sterling TR, Villarino ME, Borisov AS, Shang N, Gordin F, Bliven-Sizemore E, Hackman J, Hamilton CD, Menzies D, Kerrigan A, Weis SE, Weiner M, Wing D, Conde MB, Bozeman L, Horsburgh CR Jr, Chaisson RE; TB Trials Consortium PREVENT TB Study Team. Three months of rifapentine and isoniazid for latent tuberculosis infection. N Engl J Med. 2011 Dec 8;365(23):2155-66. doi: 10.1056/NEJMoa1104875. PMID 22150035
- [Background] Villarino ME, Scott NA, Weis SE, Weiner M, Conde MB, Jones B, Nachman S, Oliveira R, Moro RN, Shang N, Goldberg SV, Sterling TR; International Maternal Pediatric and Adolescents AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Treatment for preventing tuberculosis in children and adolescents: a randomized clinical trial of a 3-month, 12-dose regimen of a combination of rifapentine and isoniazid. JAMA Pediatr. 2015 Mar;169(3):247-55. doi: 10.1001/jamapediatrics.2014.3158. PMID 25580725